CLINICAL TRIAL: NCT00741507
Title: Unhealthy Alcohol Drinking and Anesthetic Requirement in General Anesthesia in Women
Brief Title: Unhealthy Alcohol Drinking and Anesthetic Requirement in Women
Acronym: UNADAREW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NMU-FY2008-329; NJFY-230MZ
Record Dates: First submitted 2008-08-20; First posted 2008-08-26 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: General Anesthesia
Keywords: Anesthetics; Sedatives; Analgesics
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Active Comparator): No alcohol drinking
  Interventions: Behavioral: Alcohol drinking
- 2 (Active Comparator): Mild alcohol drinking
  Interventions: Behavioral: Alcohol drinking
- 3 (Active Comparator): Moderate alcohol drinking
  Interventions: Behavioral: Alcohol drinking
- 4 (Active Comparator): Severe over alcohol drinking
  Interventions: Behavioral: Alcohol drinking
- 5 (Active Comparator): Alcohol-dependent
  Interventions: Behavioral: Alcohol drinking

INTERVENTIONS:
Behavioral: Alcohol drinking — Never drinking of alcohol
  Other Names: Ethanol use
  Arms: 1
Behavioral: Alcohol drinking — Mild drinking of alcohol assessed by "alcohol use disorders identification test (AUDIT)"
  Other Names: Ethanol use
  Arms: 2
Behavioral: Alcohol drinking — Moderate drinking of alcohol assessed by "alcohol use disorders identification test (AUDIT)"
  Other Names: Ethanol use
  Arms: 3
Behavioral: Alcohol drinking — Severe over drinking of alcohol assessed by "alcohol use disorders identification test (AUDIT)"
  Other Names: Ethanol use
  Arms: 4
Behavioral: Alcohol drinking — Alcohol-dependent assessed by "alcohol use disorders identification test (AUDIT)"
  Other Names: Ethanol use
  Arms: 5

SUMMARY:
Unhealthy alcohol drinking is negatively influencing health of people and costing a large number of annual finance via "secondhand" effects. Additionally, unhealthy alcohol use covers a spectrum that is associated with varying degrees of risk to health. The investigators hypothesized that unhealthy alcohol drinking resulted in significant increase in anesthetic requirement during general anesthesia. This investigation would clarify the association between unhealthy alcohol use and the intraoperative consumption of anesthetics, and provide clinical evidence for preoperative assessment with respect to the alcohol drinking habit.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Chinese
* 19-45yr
* Undergoing general anesthesia

Exclusion Criteria:

* A history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records.
* Participants younger than 18yr，older than 45yr or pregnancy was eliminated.
* Those who were not willing to or could not finish the whole study at any time.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Anesthetic requirements | 10 min after completion of operation

SECONDARY OUTCOMES:
Economic assessment | 1 day after operation
Odds Ratio of alcohol use and the consumption of anesthetics | 1 day after completion of study
Side effects | 30 min after completion of the study
Bispectral Index (BIS) value | 0, 5, 10, 20, 30, 45, 60, 90 min after anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China